CLINICAL TRIAL: NCT07393438
Title: Acetohydroxamic Acid Combined With a Short-Course Regimen for the Treatment of Multidrug-Resistant Tuberculosis: A Phase II Clinical Trial
Brief Title: Acetohydroxamic Acid Combined With a Short-Course Regimen for MDR-TB (AHA-PLUS)
Acronym: AHA-PLUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, yidian liu, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHA-PLUS-MDRTB-2026; 2025ZD1802404 (Other Grant/Funding Number: China National Center for Biotechnology Development)
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Multidrug-Resistant Tuberculosis; Rifampicin-resistant Tuberculosis; MDR-TB; RR-TB
Keywords: Acetohydroxamic Acid; Short-Course Regimen; BDLLfxC; BDCZ; DNA Repair; RP2D; Phase II
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — acetohydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to receive either acetohydroxamic acid plus a short-course regimen or placebo plus the same regimen, with no crossover between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors are blinded to treatment allocation. The study drug and placebo are identical in appearance, packaging, and administration schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AHA plus Short-Course Regimen (Experimental): Participants in this arm receive acetohydroxamic acid (AHA) in combination with a short-course anti-tuberculosis regimen. AHA is administered at the protocol-defined dose and schedule. All background treatments are identical to those in the control arm.
  Interventions: Drug: Acetohydroxamic Acid
- Placebo plus Short-Course Regimen (Placebo Comparator): Participants in this arm receive a matching placebo in combination with the same short-course anti-tuberculosis regimen used in the experimental arm. The placebo is identical in appearance, packaging, and administration schedule to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetohydroxamic Acid — Acetohydroxamic acid administered according to the protocol-defined dose and schedule, in combination with a short-course anti-tuberculosis regimen.
  Arms: AHA plus Short-Course Regimen
Drug: Placebo — Matching placebo identical in appearance, packaging, and administration schedule to acetohydroxamic acid, administered with the same short-course anti-tuberculosis regimen.
  Arms: Placebo plus Short-Course Regimen

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the safety, tolerability, and preliminary efficacy of acetohydroxamic acid (AHA) capsules combined with short-course regimens (BDLLfxC or BDCZ) in patients with multidrug-resistant tuberculosis (MDR-TB).

The primary objectives are to assess the safety and tolerability of AHA combined with short-course regimens, and to determine the recommended phase II dose (RP2D) of AHA.

The secondary objectives include evaluating the 8-week sputum culture conversion rate, pharmacokinetic parameters, and exploring DNA damage repair biomarkers as potential indicators of treatment response.

DETAILED DESCRIPTION:
Background:

Multidrug-resistant tuberculosis (MDR-TB) remains a significant global health challenge. Current treatment regimens face multiple bottlenecks including serious adverse effects, long treatment duration, and high cost. Acetohydroxamic acid (AHA), a urease inhibitor, represents a novel mechanism of action against tuberculosis. Recent research has revealed that Mycobacterium tuberculosis urease C (UreC) inhibits host DNA repair by interfering with the RUVBL1-RUVBL2-RAD51 complex, promoting bacterial survival. AHA, as a urease inhibitor, may block the pathogenic effect of UreC and restore host DNA repair function.

Study Design:

This is a parallel dual-study design evaluating AHA combined with two different background regimens:

* Study A: AHA + BDLLfxC regimen (6-9 months)
* Study B: AHA + BDCZ regimen (6-9 months) Each study randomizes participants in a 1:1:1:1 ratio to low-dose (500mg/day), medium-dose (750mg/day), high-dose (1000mg/day) AHA groups, or placebo group.

A double-dummy design is employed to maintain blinding, where all participants receive identical-appearing capsules regardless of treatment assignment.

The study includes a 6-9 month treatment period followed by mandatory follow-up visits at 3 and 6 months post-treatment, with optional follow-up every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to < 65 years, male or female
* Confirmed rifampicin-resistant TB (RR-TB) or multidrug-resistant TB (MDR-TB) by molecular testing (e.g., Xpert MTB/RIF) or drug susceptibility testing
* Positive sputum culture for Mycobacterium tuberculosis or positive molecular test
* Chest imaging consistent with active pulmonary TB, or histologically confirmed extrapulmonary TB (excluding CNS, osteoarticular, and disseminated TB)
* Body weight ≥ 40 kg
* Karnofsky Performance Status ≥ 50
* Adequate laboratory parameters:

  * Hemoglobin ≥ 8.0 g/dL
  * ANC ≥ 1000/mm³
  * Platelets ≥ 75,000/mm³
  * ALT/AST ≤ 3 × ULN
  * Total bilirubin ≤ 2 × ULN
  * Creatinine clearance ≥ 30 mL/min
* QTcF interval < 450 ms (male) or < 470 ms (female)
* HIV-negative, confirmed by approved testing
* No prior exposure to bedaquiline, delamanid, or linezolid for more than 1 month
* Female participants of childbearing potential must agree to use effective contraception and have a negative pregnancy test
* Signed informed consent

Exclusion Criteria:

* Central nervous system TB (e.g., TB meningitis), osteoarticular TB, or disseminated/miliary TB
* Known allergy or serious adverse reaction to any study drug or background regimen component
* Known resistance to bedaquiline, delamanid, or linezolid
* Use of anti-TB drugs within the past 30 days that may interfere with study assessments, except in documented treatment failure cases
* Severe comorbidities, including:

  * NYHA Class III-IV heart failure
  * History or risk factors for Torsades de Pointes
  * Child-Pugh B or C cirrhosis
  * Uncontrolled diabetes (HbA1c > 10%)
  * Active malignancy
* Current use of QT-prolonging medications that cannot be substituted
* Current use of MAO inhibitors or serotonergic drugs
* BMI < 17 kg/m² with severe malnutrition
* Grade 3-4 peripheral neuropathy at baseline
* Pregnant or breastfeeding women
* Any condition that, in the investigator's judgment, may interfere with study completion or data interpretation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-21 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mycobacterium tuberculosis sputum bacterial load | Baseline to Day 14
  Change in quantitative Mycobacterium tuberculosis colony-forming units (CFU) in sputum, expressed as log10 CFU/mL/day, measured using standardized microbiological culture methods.

SECONDARY OUTCOMES:
Time to sputum culture conversion | Baseline to Week 8
  Time from treatment initiation to the first of two consecutive negative Mycobacterium tuberculosis sputum cultures collected at least 24 hours apart, assessed using standardized culture methods.

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) | Baseline to Day 14
  Measurement of peak plasma concentration (Cmax) of acetohydroxamic acid using protocol-specified sampling and validated analytical methods.
Changes in inflammatory biomarkers | Baseline to Day 14
  Changes in serum inflammatory markers such as C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and other protocol-specified cytokines.
Radiographic Severity Score on Chest X-ray or CT | Baseline to Week 8
  Radiographic severity score assessed using a standardized scoring system evaluating extent of pulmonary involvement. Higher scores indicate more severe radiographic abnormalities.
Time to Peak Concentration (Tmax) | Baseline to Day 14
  Measurement of time to peak plasma concentration (Tmax) of acetohydroxamic acid based on protocol-defined pharmacokinetic sampling.
Area Under the Concentration-Time Curve (AUC) | Baseline to Day 14
  Assessment of the area under the plasma concentration-time curve (AUC) for acetohydroxamic acid using validated pharmacokinetic analysis.
Change in Cavity Size on Chest Imaging | Baseline to Week 8
  Change in the maximum diameter of pulmonary cavities measured on chest X-ray or CT using protocol-specified measurement methods.

CONTACTS AND LOCATIONS:
Overall Officials: liu yidian, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - Anhui Chest Hospital, Hefei, Anhui
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
The plan for sharing individual participant data (IPD) has not yet been finalized. Data sharing will depend on institutional policies, ethical approvals, and resource availability at the time of study completion.

REFERENCES:
- [Background] World Health Organization. Global Tuberculosis Report 2024. Geneva: WHO, 2024.
- [Background] Liu S, Guan L, Peng C, Cheng Y, Cheng H, Wang F, Ma M, Zheng R, Ji Z, Cui P, Ren Y, Li L, Shi C, Wang J, Huang X, Cai X, Qu D, Zhang H, Mao Z, Liu H, Wang P, Sha W, Yang H, Wang L, Ge B. Mycobacterium tuberculosis suppresses host DNA repair to boost its intracellular survival. Cell Host Microbe. 2023 Nov 8;31(11):1820-1836.e10. doi: 10.1016/j.chom.2023.09.010. Epub 2023 Oct 16. PMID 37848028
- [Background] Griffith DP, Gibson JR, Clinton CW, Musher DM. Acetohydroxamic acid: clinical studies of a urease inhibitor in patients with staghorn renal calculi. J Urol. 1978 Jan;119(1):9-15. doi: 10.1016/s0022-5347(17)57366-8. PMID 23442
- [Background] World Health Organization. WHO consolidated guidelines on tuberculosis. Module 4: treatment of drug-resistant tuberculosis. 2024 update. Geneva: WHO; 2024.